CLINICAL TRIAL: NCT03236623
Title: The Use of the Menthol Popsicle to Manage the Patient's Seat in the Preoperative Period: a Randomized Clinical Trial
Brief Title: Menthol Popsicle to Manage the Patient's Seat in the Preoperative Period.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Patricia Aroni, researcher, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7289
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Thirst; Perioperative Nursing
Keywords: Surgical Patient; Menthol; Clinical Study

STUDY DESIGN:
Intervention Model Description: This is a study with an experimental research design, such as a randomizedclinical trial, parallel, prospective and monocentric.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol Popsicle (Experimental): The patient will be questioned when the intensity and discomfort of thirst. After randomization, the patient assigned to the experimental group will experience a menthol popsicle. After 20 minutes of the end of the popsicle, will again be questioned as to the intensity and discomfort of thirst. The popsicle will have a support that will assist the patient in the administration of the intervention, giving him autonomy and safety in the application of the intervention.
  Interventions: Other: Menthol Popsicle
- Usual care (No Intervention): The patient will be questioned when the intensity and discomfort of thirst. After randomization, the patient assigned to the control group should receive the usual care consisting of absolute fasting the food and drinks.

INTERVENTIONS:
Other: Menthol Popsicle — The menthol popsicle composed of 0.05% menthol, 0.05% saccharin, 30ml ultrafiltered water and 2% cereal alcohol. The popsicle will have a support that will assist the patient in the administration of the intervention, giving him autonomy and safety in the application of the intervention.
  Other Names: Menthol Ice
  Arms: Menthol Popsicle

SUMMARY:
Thirst is defined as the desire to drink water. The perception and satiation of thirst constitute an interconnected network of neuronal, physiological and hormonal mechanisms that act simultaneously. In the oropharyngeal cavity are ionic channels called Transient Receptor Potential Melastatin 8 stimulated by cold temperatures and menthol, which aid in the control and decrease of the thirst intensity for providing refreshment and satiety without, however, the necessity of fluid intake In high amounts.

DETAILED DESCRIPTION:
Thus, the present study aims to: compare the intensity and discomfort of thirst in the use of the menthol popsicle and usual care in patients in the preoperative period. This is a randomized clinical trial, to be performed in a public tertiary hospital. The sample size calculation will be performed after the pilot test is conducted. Two groups will be formed through randomization. The tested intervention consists of the menthol popsicle (experimental group). The thirst intensity (primary outcome) will be measured by means of the Numerical Scale and the discomfort of thirst (secondary outcome) through the Perioperative Seat Discomfort Scale, in two moments: at the end of the first approach of the patient and 20 minutes after the intervention. The results of this research may support the decision-making of health professionals in the implementation of effective and safe actions to manage the seat of the surgical patient in the preoperative period. Another relevant aspect is the production of knowledge about the problem, which is scarce both in the national and international scenario.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Without the use of pre-anesthetic medication, until the moment of data collection;
* Conscious and alert, who recognizes himself and responds to the stimuli of the environment;
* Oriented in relation to time and space;
* Fasting for more than two hours at the time of data collection;
* Minimum time of three hours prior to the scheduled time for surgery, to approach and collect data;
* Report thirst.

Exclusion Criteria:

* Presenting a contraindication of ingestion or swallowing;
* Present mandibular trauma;
* Being nauseated or vomiting;
* Refer to allergy to mentha;
* In dialysis;
* Report sjogren's syndrome.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-11-26 (Estimated)

PRIMARY OUTCOMES:
Intensity of thirst | Measured at the beginning of the survey. For the experimental group, this measurement was measured again 20 minutes after tasting the menthol popsicle. For the control group, this measure was re-measured 20 minutes after the randomization.
  Measured from zero to ten, where zero is no thirst and ten worst thirst.
Discomfort of thirst. | Measured at the beginning of the survey. For the experimental group, this measurement was measured again 20 minutes after tasting the menthol popsicle. For the control group, this measure was re-measured 20 minutes after the randomization.
  Measured according to the Perioperative Headquarters Discomfort Scale (EDESP). The final EDESP score ranges from zero to 14 points, 14 of which correspond to the most intense discomfort related to the perioperative seat.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Aroni, Principal Investigator — University of Sao Paulo
Locations (1):
- Patricia Aroni, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No